CLINICAL TRIAL: NCT07359027
Title: Clinical Observation of Roxadustat's Effect on Anemia in Patients With Diabetic Kidney Disease (Stage III-IV)
Brief Title: Study of Roxadustat's Effect on Anemia in Patients With Diabetic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Xiangya Hospital of Central South University (Other); The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Li Xiao, professor, Second Xiangya Hospital of Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-20-20537
Record Dates: First submitted 2022-09-06; First posted 2026-01-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Kidney Disease; Anemia
MeSH Terms: conditions — Diabetic Nephropathies; Anemia | interventions — roxadustat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Roxadustat (Experimental): Oral
  Interventions: Drug: Roxadustat

INTERVENTIONS:
Drug: Roxadustat — The starting dose of Roxadustat will be defined as per the China Package Insert. The recommended starting dose of roxadustat will depend on the body weight of the patient (based on patient's empty weight prior to instillation of dialysate): 70 mg (40 to < 60 kg) tiw or 100 mg (≥ 60 kg) tiw. The frequency of hemoglobin concentration test should be ≥ once every 4 weeks. The dose will be adjusted according to the following table every 4 weeks to achieve and/or maintain hemoglobin within the target range (10.0-12.0 g/dl).
  Other Names: Roxadustat capsules

SUMMARY:
This study is a single-arm, open-label, multicenter and prospective study, which is conducted to evaluate the effect of Roxadustat on anemia in subjects with DKD (stage III-IV).

DETAILED DESCRIPTION:
This study will consist of three study periods as follows:

Screening Period: 2 weeks Treatment Period: 24weeks Follow-up Period: 4 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 60 years
2. Subject has voluntarily signed and dated an informed consent form (ICF), approved by an EC, after the nature of the study has been explained and the subject has had the opportunity to ask questions.
3. Diagnosed as Type 2 diabetic kidney disease (usually a clinical diagnosis made based on the presence of albuminuria and/or reduced eGFR in the absence of signs or symptoms of other primary causes of kidney damage), with KDOQI Stage 3 or 4 (an eGFR≧15 ml/min/1.73 m2 and <60 ml/min/1.73 m2 estimated using the CKD-EPI equation).
4. The recent Hb value during the Screening Period, must be ≥7.0 g/dL and <10 g/dL.
5. Either transferrin saturation (TSAT) ≥5% or serum ferritin ≥30 ng/mL during the screening period.
6. No use of an erythropoiesis stimulating agent for 1 week before enrolment.
7. ALT and AST ≤1.5 x ULN, and normal total bilirubin at screening visits.
8. Body weight: 40 to 100 kg inclusive.

Exclusion Criteria:

* Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

  1. Chronic kidney disease attribute to cause(s) other than diabetic kidney disease.
  2. eGFR<15ml ml/min/1.73 m2 or receiving dialysis or renal transplantation.
  3. Uncontrolled severe hypertension (SBP≧180mmHg, DBP≧100mmHg).
  4. Any clinically significant infection or evidence of an active underlying infection.
  5. New York Heart Association Class III or IV congestive heart failure.
  6. Myocardial infarction, acute coronary syndrome, stroke, seizure, or a thromboembolic event (e.g., deep venous thrombosis or pulmonary embolism) within 24 weeks prior to Day 1.
  7. Diagnosis or suspicion (e.g., complex kidney cyst of Bosniak Category IIF or higher) of renal cell carcinoma on screening renal ultrasound.
  8. History of malignancy, except the following: cancers determined to be cured or in remission for ≥5 years, curatively resected basal cell or squamous cell skin cancers, or in situ cancer at any site.
  9. Chronic inflammatory disease that could impact erythropoiesis (e.g., SLE, rheumatoid arthritis, celiac disease).
  10. Clinically significant gastrointestinal bleeding.
  11. Known history of myelodysplastic syndrome, multiple myeloma, hereditary hematologic disease such as thalassemia, sickle cell anemia, pure red cell aplasia, or other known causes for anemia other than CKD, hemosiderosis, hemochromatosis, known coagulation disorder, or hypercoagulable condition.
  12. Any prior functioning organ transplant or a scheduled organ transplantation.
  13. Anticipated elective surgery that could lead to significant blood loss during the study period.
  14. Anticipated use of dapsone or acetaminophen (paracetamol) >2.0 g/day, or >500 mg per dose repeated every 6 hours for more than 3 days.
  15. Serum albumin <2.5 g/dL.
  16. Androgen, deferoxamine, deferiprone, or deferasirox therapy within 12 weeks prior to Day 1.
  17. Life expectancy of <6 months.
  18. Blood transfusion within 12 weeks prior to Day 1 or anticipated need for transfusion.
  19. IV iron supplement during the Screening Period and /or unwilling to withhold IV iron.
  20. Immune suppressive or systemic steroid treatment within 12 weeks prior to Day 1.
  21. History of alcohol or drug abuse within the past 2 years and inability to avoid consumption of more than >3 alcoholic beverages per day.
  22. Prior treatment with any HIF-PH inhibitor (HIF-PHI).
  23. Use of an investigational medication or treatment, participation in an interventional study.
  24. Women who are pregnant or breastfeeding.
  25. Women of childbearing potential and men with sexual partners of childbearing potential who are not using adequate contraception.
  26. Any medical condition that, in the opinion of the Investigator, may pose a safety risk to a subject in this study, may confound efficacy or safety assessment, or may interfere with study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Hb level | at week 0,2,4,8,12,16,20,24
  Change in average Hb level from baseline to week 24.

SECONDARY OUTCOMES:
serum transferrin level | test at week 0,12 and 24
  Change in serum transferrin level from baseline to week 24
serum ferritin level | test at week 0,12 and 24
  Change in serum ferritin level from baseline to week 24
serum TSAT level | test at week 0,12 and 24
  Change in serum TSAT level from baseline to week 24
serum iron level | test at week 0,12 and 24
  Change in serum iron level from baseline to week 24
FPG and PPG | test at week 0,12 and 24
  Change in FPG and PPG levels from baseline to week 24
HbA1C level | test at week 0,12 and 24
  Change in HbA1C level from baseline to week 24
Triglycerides, Cholesterol, HDL, LDL levels | test at week 0,12 and 24
  Change in triglycerides, cholesterol, HDL, and LDL levels from baseline to week 24
apolipoprotein level | test at week 0,12 and 24
  Change in apolipoprotein level from baseline to week 24
Physical parameters | test at week 0,12 and 24
  SF-36 summary scores (PCS and MCS), physical functioning and vitality

OTHER OUTCOMES:
UACR | test at week 0,2,4,8,12,16,20,24
  Change in UACR level from baseline to week 24
serum creatinine | test at week 0,2,4,8,12,16,20,24
  Change in serum creatinine level from baseline to week 24
uric acid | test at week 0,2,4,8,12,16,20,24
  Change in uric acid level from baseline to week 24
eGFR | test at week 0,2,4,8,12,16,20,24
  Change in eGFR from baseline to week 24
urine-NGAL | test at week 0,24
  Change in urine-NGAL level from baseline to week 24
24h-urinalysis | test at week 0,24
  Change in 24h-urinalysis from baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Lin Sun, doctor, Principal Investigator — Department of Nephrology, Second Xiangya hospital of central south university, Changsha, China.
Locations (1):
- Second Xiangya Hospital, Central South University, Changsha, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen N, Hao C, Peng X, Lin H, Yin A, Hao L, Tao Y, Liang X, Liu Z, Xing C, Chen J, Luo L, Zuo L, Liao Y, Liu BC, Leong R, Wang C, Liu C, Neff T, Szczech L, Yu KP. Roxadustat for Anemia in Patients with Kidney Disease Not Receiving Dialysis. N Engl J Med. 2019 Sep 12;381(11):1001-1010. doi: 10.1056/NEJMoa1813599. Epub 2019 Jul 24. PMID 31340089
- [Background] Chen N, Hao C, Liu BC, Lin H, Wang C, Xing C, Liang X, Jiang G, Liu Z, Li X, Zuo L, Luo L, Wang J, Zhao MH, Liu Z, Cai GY, Hao L, Leong R, Wang C, Liu C, Neff T, Szczech L, Yu KP. Roxadustat Treatment for Anemia in Patients Undergoing Long-Term Dialysis. N Engl J Med. 2019 Sep 12;381(11):1011-1022. doi: 10.1056/NEJMoa1901713. Epub 2019 Jul 24. PMID 31340116
- [Background] Yan Z, Xu G. A Novel Choice to Correct Inflammation-Induced Anemia in CKD: Oral Hypoxia-Inducible Factor Prolyl Hydroxylase Inhibitor Roxadustat. Front Med (Lausanne). 2020 Aug 6;7:393. doi: 10.3389/fmed.2020.00393. eCollection 2020. PMID 32850902